CLINICAL TRIAL: NCT05652452
Title: Neurodynamic Sliders Promote Flexibility in Tight Hamstring Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B670201630354
Record Dates: First submitted 2018-07-04; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Hamstring Injury; Neurodynamics; Range of Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodynamics (Experimental)
  Interventions: Other: Neurodynamics
- Static stretch (Active Comparator)
  Interventions: Other: Static stretch

INTERVENTIONS:
Other: Neurodynamics — Subjects in the neurodynamic group performed the 'Seated Straight Leg Slider' (SSLS) (Fig.1). To execute this sliding technique, subjects assumed a seated slump position (thoracic and lumbar flexion) which they needed to maintain throughout the exercise. This SSLS consisted of alternating movements towards knee extension and ankle dorsiflexion (increase of neural tension) combined with cervical extension (decrease of neural tension) on one hand, and knee flexion and ankle plantar flexion (decrease neural tension) combined with cervical flexion (increase of neural tension) on the other. During this 6-week period, each subject in this neurodynamic slider group was instructed to perform 3 sets of 20 repetitions on a daily basis for 6 weeks.
  Arms: Neurodynamics
Other: Static stretch — Subjects in the control group were instructed to perform a standard standing static stretch with the heel of the dominant leg taking support on a chair. Then they had to move the pelvis into anteversion, simultaneously inducing a forward lean of the trunk, until the clear sensation of hamstring stretch was perceived at the posterior aspect of the thigh. Again, the execution of the exercise was thoroughly explained and evaluated by the researchers and subjects sent home with a comprehensive instruction guide and supporting pictures. Each subject was instructed to do 3 repetitions of 30 second static stretches on a daily basis during the 6-week intervention.
  Arms: Static stretch

SUMMARY:
The goal of this study is to explore the intervention effect of home-based neurodynamic slider program on hamstring flexibility. Fifty physically active male subjects will be randomly assigned to either performing a neurodynamic sliding technique (3x20 reps) or a static stretching protocol (3x30") on a daily basis for a 6-week period. Hamstring flexibility will be assessed by means of the Straight Leg Raise at baseline, immediately after the intervention and after 4 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* male
* aged between 18-30yrs
* recreationally/competitively active
* limited hamstring flexibility (Tight Hamstring Syndrome) (SLR≤75°)

Exclusion Criteria:

* a history of any musculotendinous hamstring injury in the previous year
* a history of neurological or orthopedic disorder affecting the lower extremities
* a history of lumbar disc herniation; or (4) a history of a cervical whiplash injury

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Hamstring flexibility | at Baseline
  Straight leg raise by means of an app based goniometer
Hamstring flexibility | 6 weeks after intervention
  Straight leg raise by means of an app based goniometer
Hamstring flexibility | 4 weeks after retention period
  Straight leg raise by means of an app based goniometer

IPD SHARING:
Plan to Share IPD: No